CLINICAL TRIAL: NCT00970593
Title: A RANDOMIZED, PARALLEL-GROUP, OPEN-LABEL, PLACEBO CONTROLLED STUDY OF THE EFFECT OF OAP-189 ON THE PHARMACOKINETICS AND PHARMACODYNAMICS OF METFORMIN IN DIABETIC SUBJECTS.
Brief Title: Study Evaluating Safety, Tolerability, And Action Of OAP-189 In Subjects With Type 2 Diabetes On Metformin
Acronym: 3283K1-1008-US
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3283K1-1008; B2201004 (Other: Alias Study Number)
Record Dates: First submitted 2009-09-01; First posted 2009-09-02 (Estimated); Results first posted 2020-11-02 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- OAP-189 (Placebo Comparator)
  Interventions: Drug: OAP-189
- 2 (Placebo Comparator)
  Interventions: Drug: placebo comparator

INTERVENTIONS:
Drug: OAP-189 — Group 1: OAP-189 BID (0.2 mg BID) x 7 days Group 2: OAP-189 (0.4 mg BID) x 7 days Group 3: OAP-189 QD (0.9 mg x 7 days followed by 1.2 mg x 7 days; MR formulation) Group 4: OAP-189 QD (1.2 mg x 7 days followed by 1.6 mg x 7 days; MR formulation) Group 5: OAP-189 QD (1.2 mg x 7 days followed by 1.6 mg x 7 days; different MR formulation) Group 6: OAP-189 QD (1.2 mg x 7 days followed by 1.6 mg x 7 days; different MR formulation)
  Arms: OAP-189
Drug: placebo comparator — Group 1 & 2: PBO x 7 days BID Group 3: PBO QD x 14 days Group 4: PBO QD x 14 days Group 5: PBO QD x 14 days Group 6: PBO QD x 14 days
  Arms: 2

SUMMARY:
This is a study to evaluate the safety, tolerability, and activity of OAP-189 in subjects with type 2 diabetes who are taking metformin for their diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have been diagnosed with type 2 diabetes, with HbA1c level >=7.0% and <=11.0% and a fasting glucose level <=280 mg/dL.
* Men or women of nonchildbearing potential (WONCBP), aged 18 to 65 years inclusive on study day 1.
* Body mass index in the range of 27 to 40kg/m² (inclusive) and body weight >=50 kg.
* Subjects must be otherwise generally healthy, but may be enrolled with a stable chronic illness, if it is well controlled and does not interfere with the primary objective of the study.
* Subjects must currently be treated for diabetes with metformin alone at a total daily dose of >=1gm (administered QD or BID) and that dose must have been stable for at least 4 weeks before study day 1.
* Nonsmoker.

Exclusion Criteria:

* Any significant disease with the exception of diabetes mellitus.
* Any surgical or medical condition that may interfere with the absorption, distribution, metabolism, or excretion of the investigational product.
* Acute disease state (eg, nausea, vomiting, fever, or diarrhea) within 7 days before study day 1.
* Any clinically important problems in physical examination results, vitals sign measurements, ECGs, or clinical laboratory test results.
* Positive serologic findings for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg), and/or hepatitis C virus (HCV) antibodies.
* Positive findings of urine drug screen
* Use of any investigational or non-permitted prescription drug within 30 days before investigational product administration.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2009-09-02 (Actual); Primary Completion 2011-07-25 (Actual); Study Completion 2011-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Profil Institute for Clincal Research, Chula Vista, California
  - Cetero Research - Miami, Miami Gardens, Florida

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3283K1-1008&StudyName=Study%20Evaluating%20Safety%2C%20Tolerability%2C%20And%20Action%20Of%20OAP-189%20In%20Subjects%20With%20Type%202%20Diabetes%20On%20Metformin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants received the background metformin immediate release tablets, during the 4 weeks run-in period. Compliant participants were then randomized to study treatments for a maximum period of 31 days.
Groups:
- OAP-189 0.2 mg IR: Participants received OAP-189 0.2 milligram (mg), immediate release (IR) infusion subcutaneously twice daily from Day 1 to Day 7 along with background metformin 850 mg immediate release tablets or as per standard clinical practice (based on the dose prior to randomization).
- OAP-189 0.4 mg IR: Participants received OAP-189 0.4 mg, IR infusion subcutaneously twice daily from Day 1 to Day 7 along with background metformin 850 mg immediate release tablets or as per standard clinical practice (based on the dose prior to randomization).
- OAP-189 MR (0.05:1 Z/P Ratio) 0.9 mg Followed by 1.2 mg: Participants received OAP-189 0.9 mg, modified release (MR) infusion (with 0.05:1 zinc to peptide [Z/P] ratio) subcutaneously once daily from Day 1 to Day 7 followed by OAP-189 1.2 mg, MR infusion subcutaneously once daily from Day 8 to Day 14 along with background metformin 850 mg immediate release tablets or as per standard clinical practice (based on the dose prior to randomization).
- OAP-189 MR (0.1:1 Z/P Ratio) 1.2 mg Followed by 1.6 mg: Participants received OAP-189 1.2 mg, MR infusion (with 0.1:1 Z/P ratio) subcutaneously once daily from Day 1 to Day 7 followed by OAP-189 1.6 mg, MR infusion subcutaneously once daily from Day 8 to Day 14 along with background metformin 850 mg immediate release tablets or as per standard clinical practice (based on the dose prior to randomization).
- OAP-189 MR (0.25:1 Z/P Ratio) 1.2 mg Followed by 1.6 mg: Participants received OAP-189 1.2 mg, MR infusion (with 0.25:1 Z/P ratio) subcutaneously once daily from Day 1 to Day 7 followed by OAP-189 1.6 mg, MR infusion subcutaneously once daily from Day 8 to Day 14 along with background metformin 850 mg immediate release tablets or as per standard clinical practice (based on the dose prior to randomization).
- Placebo IR: Participants received placebo matched to OAP-189, IR infusion subcutaneously twice daily from Day 1 to Day 7 along with background metformin 850 mg immediate release tablets or as per standard clinical practice (based on the dose prior to randomization).
- Placebo MR: Participants received placebo matched to OAP-189, MR infusion subcutaneously once daily from Day 1 to Day 14 along with background metformin 850 mg immediate release tablets or as per standard clinical practice (based on the dose prior to randomization).
Period: Overall Study
Arm/Group | OAP-189 0.2 mg IR | OAP-189 0.4 mg IR | OAP-189 MR (0.05:1 Z/P Ratio) 0.9 mg Followed by 1.2 mg | OAP-189 MR (0.1:1 Z/P Ratio) 1.2 mg Followed by 1.6 mg | OAP-189 MR (0.25:1 Z/P Ratio) 1.2 mg Followed by 1.6 mg | Placebo IR | Placebo MR
Started | 11 | 15 | 13 | 12 | 20 | 5 | 16
Completed | 10 | 14 | 7 | 12 | 20 | 5 | 14
Not Completed | 1 | 1 | 6 | 0 | 0 | 0 | 2
Not completed — Adverse Event | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Discontinuation of study by sponsor | 0 | 0 | 5 | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all randomly assigned participants who received at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | OAP-189 0.2 mg IR | OAP-189 0.4 mg IR | OAP-189 MR (0.05:1 Z/P Ratio) 0.9 mg Followed by 1.2 mg | OAP-189 MR (0.1:1 Z/P Ratio) 1.2 mg Followed by 1.6 mg | OAP-189 MR (0.25:1 Z/P Ratio) 1.2 mg Followed by 1.6 mg | Placebo IR | Placebo MR | Total
Number analyzed (Participants) | 11 | 15 | 13 | 12 | 20 | 5 | 16 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.00 (8.65) | 53.60 (6.33) | 52.69 (3.12) | 54.92 (6.69) | 51.50 (9.64) | 53.80 (9.34) | 54.75 (6.83) | 53.57 (7.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 3 | 4 | 4 | 2 | 6 | 26
  Male | 8 | 11 | 10 | 8 | 16 | 3 | 10 | 66

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinically Significant Physical Examination Abnormalities
Description: Physical examination included examination of skin, head, eyes, ears, nose, throat (HEENT), heart, lungs, abdomen, extremities, neurological function, back and lymph nodes. Clinically significant physical examination abnormalities were considered as adverse events based on investigator's discretion.
Time Frame: Baseline up to 17 days after last dose of study drug (Day 31)
Population: Safety population included all randomly assigned participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Groups:
- OAP-189 0.2 mg IR: Participants received OAP-189 0.2 mg, IR infusion subcutaneously twice daily from Day 1 to Day 7 along with background metformin 850 mg immediate release tablets or as per standard clinical practice (based on the dose prior to randomization).
- OAP-189 MR (0.05:1 Z/P Ratio) 0.9 mg Followed by 1.2 mg: Participants received OAP-189 0.9 mg, MR infusion (with 0.05:1 zinc to peptide [Z/P] ratio) subcutaneously once daily from Day 1 to Day 7 followed by OAP-189 1.2 mg, MR infusion subcutaneously once daily from Day 8 to Day 14 along with background metformin 850 mg immediate release tablets or as per standard clinical practice (based on the dose prior to randomization).
Arm/Group | OAP-189 0.2 mg IR | OAP-189 0.4 mg IR | OAP-189 MR (0.05:1 Z/P Ratio) 0.9 mg Followed by 1.2 mg | OAP-189 MR (0.1:1 Z/P Ratio) 1.2 mg Followed by 1.6 mg | OAP-189 MR (0.25:1 Z/P Ratio) 1.2 mg Followed by 1.6 mg | Placebo IR | Placebo MR
Number analyzed (Participants) | 11 | 15 | 13 | 12 | 20 | 5 | 16
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Clinically Significant Vital Signs Abnormalities
Description: Criteria for clinically significant vital sign abnormalities: sitting systolic blood pressure (SBP) of (greater than equal to) >=160 millimeter of mercury (mmHg), (less than equal to) <=90 mmHg, >=20 mmHg increase and decrease from baseline; sitting diastolic blood pressure (DBP) of >=100 mmHg, <=50 mmHg, >=15 mmHg increase and decrease from baseline; heart rate of >=120 beats per minute (bpm), <=45 bpm, (greater than) >15 bpm increase and decrease from baseline, orthostatic SBP: decrease of >=20 mm Hg from sitting value, orthostatic DBP: decrease of >=20 mm Hg from sitting value, orthostatic heart rate: increase of >=30 bpm from sitting value, oral temperature of (less than) <35 or >38.3 degree celsius, respiratory rate of <10 or >25 breaths per minute, weight: maximum increase or decrease of >=7 percent (%) from baseline.
Time Frame: Baseline up to 17 days after last dose of study drug (Day 31)
Population: Safety population included all randomly assigned participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | OAP-189 0.2 mg IR | OAP-189 0.4 mg IR | OAP-189 MR (0.05:1 Z/P Ratio) 0.9 mg Followed by 1.2 mg | OAP-189 MR (0.1:1 Z/P Ratio) 1.2 mg Followed by 1.6 mg | OAP-189 MR (0.25:1 Z/P Ratio) 1.2 mg Followed by 1.6 mg | Placebo IR | Placebo MR
Number analyzed (Participants) | 11 | 15 | 13 | 12 | 20 | 5 | 16
participants | 1 | 2 | 1 | 2 | 4 | 0 | 1

3. Primary Outcome: Number of Participants With Clinically Significant 12-Lead Electrocardiogram (ECG) Abnormalities
Description: Criteria for clinically significant ECG abnormalities: PR interval >=220 millisecond (msec) or a change of >=20 msec from baseline values, QRS interval >=120 msec, QTc interval >450 msec (in males) and >470 msec (in females).
Time Frame: Baseline up to 17 days after last dose of study drug (Day 31)
Population: Safety population included all randomly assigned participants who received at least 1 dose of study medication. Here, 'N' (Number of Participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Number; unit: participants
Arm/Group | OAP-189 0.2 mg IR | OAP-189 0.4 mg IR | OAP-189 MR (0.05:1 Z/P Ratio) 0.9 mg Followed by 1.2 mg | OAP-189 MR (0.1:1 Z/P Ratio) 1.2 mg Followed by 1.6 mg | OAP-189 MR (0.25:1 Z/P Ratio) 1.2 mg Followed by 1.6 mg | Placebo IR | Placebo MR
Number analyzed (Participants) | 11 | 15 | 8 | 12 | 20 | 5 | 14
participants | 0 | 0 | 2 | 4 | 4 | 0 | 7

4. Primary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities
Description: Hematocrit, haemoglobin: decrease of >=0.05 L/L and >=20 g/L from baseline respectively, WBC count:<3*10^9 /L, neutrophils: <1.5*10^9 /L, platelet count: <100*10^9 /L, eosinophil: <0.5*10^9 /L; prothrombin time, partial thromboplastin time >1.5*upper limit of normal (ULN); sodium:>5 mmol/L above ULN or below lower limit of normal(LLN), potassium >0.5 mmol/L above ULN or below LLN, creatinine >1.36*ULN, blood urea nitrogen >1.5*ULN, glucose (fasting) >0.83 mmol/L above ULN or below LLN, glucose (non-fasting) >5 mmol/L above ULN or >0.56 below LLN, calcium, magnesium: Change of >=0.25 and >=0.21 mmol/L from baseline respectively, phosphorus >0.162 mmol/L above ULN or below LLN, total protein, albumin, uric acid: change of >=20g/L, >=10 g/L, >0.119 mmol/L from baseline respectively, creatinine kinase >3*ULN, total cholesterol >7.77 mmol/L, triglycerides >3.39 mmol/L: AST, ALT, total bilirubin >2*ULN, alkaline phosphatase >1.5*ULN, alpha-glumatyl transferase, lactate dehydrogenase >3*ULN.
Time Frame: Baseline up to 17 days after last dose of study drug (Day 31)
Population: Safety population included all randomly assigned participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | OAP-189 0.2 mg IR | OAP-189 0.4 mg IR | OAP-189 MR (0.05:1 Z/P Ratio) 0.9 mg Followed by 1.2 mg | OAP-189 MR (0.1:1 Z/P Ratio) 1.2 mg Followed by 1.6 mg | OAP-189 MR (0.25:1 Z/P Ratio) 1.2 mg Followed by 1.6 mg | Placebo IR | Placebo MR
Number analyzed (Participants) | 11 | 15 | 13 | 12 | 20 | 5 | 16
participants | 10 | 15 | 13 | 9 | 19 | 5 | 15

5. Primary Outcome: Number of Participants With Injection Site Reactions
Description: Injection site reactions included irritation, erythema, pain, hematoma, inflammation.
Time Frame: Baseline up to 17 days after last dose of study drug (Day 31)
Population: Safety population included all randomly assigned participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | OAP-189 0.2 mg IR | OAP-189 0.4 mg IR | OAP-189 MR (0.05:1 Z/P Ratio) 0.9 mg Followed by 1.2 mg | OAP-189 MR (0.1:1 Z/P Ratio) 1.2 mg Followed by 1.6 mg | OAP-189 MR (0.25:1 Z/P Ratio) 1.2 mg Followed by 1.6 mg | Placebo IR | Placebo MR
Number analyzed (Participants) | 11 | 15 | 13 | 12 | 20 | 5 | 16
participants
  Irritation | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Erythema | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Pain | 0 | 0 | 0 | 2 | 1 | 0 | 0
  Hematoma | 0 | 0 | 0 | 0 | 3 | 0 | 1
  Inflammation | 0 | 0 | 0 | 0 | 0 | 0 | 1

6. Primary Outcome: Number of Participants With Clinically Significant Fasting Glucose Level Abnormalities
Description: Criteria: Blood glucose levels >15 milligram per deciliter (mg/dL) above ULN or >15 mg/dL below LLN.
Time Frame: Baseline up to 17 days after last dose of study drug (Day 31)
Population: Safety population included all randomly assigned participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | OAP-189 0.2 mg IR | OAP-189 0.4 mg IR | OAP-189 MR (0.05:1 Z/P Ratio) 0.9 mg Followed by 1.2 mg | OAP-189 MR (0.1:1 Z/P Ratio) 1.2 mg Followed by 1.6 mg | OAP-189 MR (0.25:1 Z/P Ratio) 1.2 mg Followed by 1.6 mg | Placebo IR | Placebo MR
Number analyzed (Participants) | 11 | 15 | 13 | 12 | 20 | 5 | 16
participants | 10 | 15 | 13 | 9 | 19 | 5 | 15

7. Primary Outcome: Number of Participants With Hypoglycaemia
Description: Hypoglycaemia is a condition characterized by abnormally low blood glucose (blood sugar) levels, usually <=50 mg/dL.
Time Frame: Baseline up to 17 days after last dose of study drug (Day 31)
Population: Safety population included all randomly assigned participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | OAP-189 0.2 mg IR | OAP-189 0.4 mg IR | OAP-189 MR (0.05:1 Z/P Ratio) 0.9 mg Followed by 1.2 mg | OAP-189 MR (0.1:1 Z/P Ratio) 1.2 mg Followed by 1.6 mg | OAP-189 MR (0.25:1 Z/P Ratio) 1.2 mg Followed by 1.6 mg | Placebo IR | Placebo MR
Number analyzed (Participants) | 11 | 15 | 13 | 12 | 20 | 5 | 16
participants | 0 | 0 | 0 | 2 | 1 | 0 | 0

8. Primary Outcome: Number of Participants With Drug-Induced Liver Injury
Description: Criteria for drug induced liver injury: Levels of aspartate transaminase (AST) or alanine transaminase (ALT) should be >= 3 times ULN concurrent with a total bilirubin of >=2 times ULN with no evidence of hemolysis and an alkaline phosphatase should be <=2 times ULN.
Time Frame: Baseline up to 17 days after last dose of study drug (Day 31)
Population: Safety population included all randomly assigned participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | OAP-189 0.2 mg IR | OAP-189 0.4 mg IR | OAP-189 MR (0.05:1 Z/P Ratio) 0.9 mg Followed by 1.2 mg | OAP-189 MR (0.1:1 Z/P Ratio) 1.2 mg Followed by 1.6 mg | OAP-189 MR (0.25:1 Z/P Ratio) 1.2 mg Followed by 1.6 mg | Placebo IR | Placebo MR
Number analyzed (Participants) | 11 | 15 | 13 | 12 | 20 | 5 | 16
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Primary Outcome: Change From Baseline in Predose Fasting Glucose Levels at Day 8
Description: Fasting glucose levels were determined before administration of OAP-189 using a glucometer.
Time Frame: Baseline, Day 8
Population: Safety population included all randomly assigned participants who received at least 1 dose of study medication. Here, 'n' signifies those participants who were evaluable at specified time points. This outcome measure was not to be analyzed in participants of OAP-189 0.2, 0.4 mg IR and Placebo IR as pre-specified in the protocol.
Measure: Mean (Standard Deviation); unit: millimole per liter
Arm/Group | OAP-189 MR (0.05:1 Z/P Ratio) 0.9 mg Followed by 1.2 mg | OAP-189 MR (0.1:1 Z/P Ratio) 1.2 mg Followed by 1.6 mg | OAP-189 MR (0.25:1 Z/P Ratio) 1.2 mg Followed by 1.6 mg | Placebo MR
Number analyzed (Participants) | 13 | 12 | 20 | 16
millimole per liter
  Baseline: number analyzed (Participants) | 12 | 12 | 20 | 16
  Baseline | 10.02 (2.373) | 10.06 (2.583) | 9.27 (2.148) | 9.01 (1.769)
  Change at Day 8: number analyzed (Participants) | 11 | 10 | 20 | 12
  Change at Day 8 | -1.37 (2.222) | -2.75 (1.663) | -2.47 (1.400) | -0.25 (1.166)
Statistical Analysis 1: Comparison: OAP-189 MR (0.05:1 Z/P Ratio) 0.9 mg Followed by 1.2 mg vs Placebo MR; The Mixed model used fixed effects of treatment, study day and treatment by study day interaction; Test type: Superiority or Other; LS mean difference = -0.75, 95% CI 2-sided [-1.79 to 0.29], Standard Error of Mean 0.526
Statistical Analysis 2: Comparison: OAP-189 MR (0.1:1 Z/P Ratio) 1.2 mg Followed by 1.6 mg vs Placebo MR; The Mixed model used fixed effects of treatment, study day and treatment by study day interaction; Test type: Superiority or Other; LS mean difference = -1.90, 95% CI 2-sided [-2.98 to -0.83], Standard Error of Mean 0.543
Statistical Analysis 3: Comparison: OAP-189 MR (0.25:1 Z/P Ratio) 1.2 mg Followed by 1.6 mg vs Placebo MR; The Mixed model used fixed effects of treatment, study day and treatment by study day interaction; Test type: Superiority or Other; LS mean difference = -2.15, 95% CI 2-sided [-3.06 to -1.24], Standard Error of Mean 0.458

10. Primary Outcome: Change From Baseline in Predose Fasting Glucose Levels at Day 15
Description: Fasting glucose levels were determined before administration of OAP-189 using a glucometer.
Time Frame: Baseline, Day 15
Population: Safety population included all randomly assigned participants who received at least 1 dose of study medication. Here, 'N' signifies those participants who were evaluable for this measure. This outcome measure was not to be analyzed in participants of OAP-189 0.2, 0.4 mg IR and Placebo IR as pre-specified in protocol.
Measure: Mean (Standard Deviation); unit: millimole per liter
Arm/Group | OAP-189 MR (0.05:1 Z/P Ratio) 0.9 mg Followed by 1.2 mg | OAP-189 MR (0.1:1 Z/P Ratio) 1.2 mg Followed by 1.6 mg | OAP-189 MR (0.25:1 Z/P Ratio) 1.2 mg Followed by 1.6 mg | Placebo MR
Number analyzed (Participants) | 7 | 12 | 20 | 14
millimole per liter | -2.62 (0.998) | -3.87 (1.783) | -3.49 (1.643) | -0.33 (1.273)
Statistical Analysis 1: Comparison: OAP-189 MR (0.05:1 Z/P Ratio) 0.9 mg Followed by 1.2 mg vs Placebo MR; The Mixed model used fixed effects of treatment, study day and treatment by study day interaction; Test type: Superiority or Other; LS Mean difference = -2.37, 95% CI 2-sided [-3.52 to -1.22], Standard Error of Mean 0.580
Statistical Analysis 2: Comparison: OAP-189 MR (0.1:1 Z/P Ratio) 1.2 mg Followed by 1.6 mg vs Placebo MR; The Mixed model used fixed effects of treatment, study day and treatment by study day interaction; Test type: Superiority or Other; LS mean difference = -3.18, 95% CI 2-sided [-4.16 to -2.20], Standard Error of Mean 0.495
Statistical Analysis 3: Comparison: OAP-189 MR (0.25:1 Z/P Ratio) 1.2 mg Followed by 1.6 mg vs Placebo MR; The Mixed model used fixed effects of treatment, study day and treatment by study day interaction; Test type: Superiority or Other; LS mean difference = -3.14, 95% CI 2-sided [-4.01 to -2.28], Standard Error of Mean 0.437

11. Other Pre Specified Outcome: Plasma Concentration Versus Time Summary of Metformin Following Single Dose of OAP-189
Description: Concentration versus time summary was calculated by setting concentration values below the lower limit of quantification (LLOQ =2 nanogram per millliter) to zero. Summary statistics were not to be presented if number of observations above lower limit of quantification (NALQ) =0.
Time Frame: Pre-dose (2 hours before dosing), 1, 2, 3, 4, 6 hours post-dose on Day 14
Population: Pharmacokinetic (PK) analysis set. Here, 'N' (Number of Participants analyzed) signifies those participants who were evaluable for this measure. This outcome measure was not to be analyzed in participants of OAP-189 0.2, 0.4 mg IR, Placebo IR, OAP-189 MR (0.25:1 Z/P ratio) 1.2 mg followed by 1.6 mg and Placebo MR as pre-specified in protocol.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Arm/Group | OAP-189 MR (0.05:1 Z/P Ratio) 0.9 mg Followed by 1.2 mg | OAP-189 MR (0.1:1 Z/P Ratio) 1.2 mg Followed by 1.6 mg
Number analyzed (Participants) | 7 | 12
nanogram per milliliter
  Pre-dose | 318.7 (140.36) | 455.6 (246.43)
  1 hour post dose | 899.1 (344.02) | 990.9 (453.01)
  2 hour post dose | 885.4 (364.20) | 1112 (652.61)
  3 hour post dose | 881.4 (357.83) | 1063 (613.86)
  4 hour post dose | 912.3 (381.22) | 943.7 (474.35)
  6 hour post dose | 869.7 (215.27) | 804.8 (349.20)

12. Other Pre Specified Outcome: Plasma Concentration Versus Time Summary of Metformin Following Multiple Dose of OAP-189
Description: as for outcome 11
Time Frame: Pre-dose (2 hours before dosing), 1, 2, 3, 4, 6, 8, 10, 12, 14, 16, 24 hours post-dose on Day 7
Population: PK analysis set. Here, 'N' = participants evaluable for this measure. This outcome was not to be analyzed in participants of Placebo IR, OAP-189 MR (0.05:1 Z/P ratio) 0.9 mg followed by 1.2 mg, OAP-189 MR (0.1:1 Z/P ratio) 1.2 mg followed by 1.6 mg, OAP-189 MR (0.25:1 Z/P ratio) 1.2 mg followed by 1.6 mg and Placebo MR as pre-specified in protocol.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Arm/Group | OAP-189 0.2 mg IR | OAP-189 0.4 mg IR
Number analyzed (Participants) | 10 | 14
nanogram per milliliter
  Pre-dose | 544.7 (334.72) | 558.9 (386.19)
  1 hour post dose | 998.8 (360.42) | 1276 (858.80)
  2 hour post dose | 980.7 (336.37) | 1084 (582.26)
  3 hour post dose | 995.8 (342.21) | 985.5 (424.50)
  4 hour post dose | 938.3 (355.38) | 974.7 (504.81)
  6 hour post dose | 804.6 (343.23) | 854.0 (415.21)
  8 hour post dose | 617.0 (265.18) | 735.4 (350.03)
  10 hour post dose | 462.4 (194.50) | 658.1 (457.83)
  12 hour post dose | 987.2 (442.22) | 1029 (477.30)
  14 hour post dose | 972.6 (415.05) | 976.4 (497.10)
  16 hour post dose | 889.7 (465.26) | 906.1 (418.88)
  24 hour post dose | 455.1 (488.53) | 503.5 (334.27)

13. Other Pre Specified Outcome: Plasma Concentration Versus Time Summary of Single Dose of OAP-189
Description: Concentration versus time summary was calculated by setting concentration values below the lower limit of quantification (LLOQ = 0.500 nanogram per millliter) to zero. Summary statistics were not to be presented if number of observations above lower limit of quantification (NALQ) =0.
Time Frame: Pre-dose (2 hours before dosing), 2, 4, 6 hours post-dose on Day 7; Pre-dose (2 hours before dosing), 1, 2, 3, 4, 6, 8, 10, 12, 14, 16, 24, 48, 72 hours post-dose on Day 14
Population: PK analysis set. Here, 'n' signifies those participants who were evaluable at specified time points. This outcome measure was not to be analyzed in participants of OAP-189 0.2, 0.4 mg IR, Placebo IR and MR as pre-specified in protocol.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Arm/Group | OAP-189 MR (0.05:1 Z/P Ratio) 0.9 mg Followed by 1.2 mg | OAP-189 MR (0.1:1 Z/P Ratio) 1.2 mg Followed by 1.6 mg | OAP-189 MR (0.25:1 Z/P Ratio) 1.2 mg Followed by 1.6 mg
Number analyzed (Participants) | 13 | 12 | 20
nanogram per milliliter
  Day 7: Pre-dose: number analyzed (Participants) | 12 | 12 | 20
  Day 7: Pre-dose | 2.173 (0.55480) | 3.253 (1.2371) | 2.313 (1.0927)
  Day 7: 2 hour post dose: number analyzed (Participants) | 12 | 12 | 20
  Day 7: 2 hour post dose | 8.065 (2.8023) | 11.56 (8.9549) | 5.380 (3.2235)
  Day 7: 4 hour post dose: number analyzed (Participants) | 12 | 12 | 20
  Day 7: 4 hour post dose | 10.40 (4.8907) | 14.21 (10.429) | 6.113 (2.8196)
  Day 7: 6 hour post dose: number analyzed (Participants) | 12 | 12 | 20
  Day 7: 6 hour post dose | 9.173 (4.4176) | 11.71 (6.7732) | 5.249 (2.7225)
  Day 14: Pre-dose: number analyzed (Participants) | 7 | 12 | 20
  Day 14: Pre-dose | 3.350 (0.85499) | 4.550 (2.0888) | 3.404 (1.6691)
  Day 14: 1 hour post dose: number analyzed (Participants) | 7 | 12 | 20
  Day 14: 1 hour post dose | 6.740 (3.4367) | 18.46 (34.903) | 7.686 (5.0265)
  Day 14: 2 hour post dose: number analyzed (Participants) | 7 | 12 | 20
  Day 14: 2 hour post dose | 9.747 (4.8634) | 19.53 (23.410) | 8.492 (4.0211)
  Day 14: 3 hour post dose: number analyzed (Participants) | 7 | 12 | 20
  Day 14: 3 hour post dose | 11.23 (4.4618) | 19.79 (17.035) | 8.969 (3.6809)
  Day 14: 4 hour post dose: number analyzed (Participants) | 7 | 12 | 20
  Day 14: 4 hour post dose | 11.70 (4.4452) | 17.88 (12.785) | 8.911 (3.5977)
  Day 14: 6 hour post dose: number analyzed (Participants) | 7 | 12 | 20
  Day 14: 6 hour post dose | 9.611 (3.7471) | 14.97 (10.234) | 7.353 (3.2211)
  Day 14: 8 hour post dose: number analyzed (Participants) | 7 | 12 | 20
  Day 14: 8 hour post dose | 8.094 (3.3158) | 12.83 (7.6125) | 6.326 (2.7418)
  Day 14: 10 hour post dose (: number analyzed (Participants) | 7 | 12 | 20
  Day 14: 10 hour post dose ( | 6.991 (2.6902) | 10.13 (5.8597) | 5.845 (2.1174)
  Day 14: 12 hour post dose: number analyzed (Participants) | 7 | 12 | 20
  Day 14: 12 hour post dose | 5.431 (2.0067) | 7.939 (4.6575) | 5.152 (2.3713)
  Day 14: 14 hour post dose: number analyzed (Participants) | 7 | 12 | 20
  Day 14: 14 hour post dose | 4.341 (1.5433) | 6.708 (3.4394) | 4.604 (1.7001)
  Day 14: 16 hour post dose: number analyzed (Participants) | 7 | 12 | 20
  Day 14: 16 hour post dose | 4.160 (0.93113) | 5.993 (3.0649) | 4.612 (1.8386)
  Day 14: 24 hour post dose: number analyzed (Participants) | 7 | 12 | 20
  Day 14: 24 hour post dose | 2.910 (0.70512) | 3.911 (1.7983) | 3.688 (1.2721)
  Day 14: 48 hour post dose: number analyzed (Participants) | 7 | 12 | 20
  Day 14: 48 hour post dose | 1.285 (0.29853) | 1.781 (1.1929) | 1.968 (1.1127)
  Day 14: 72 hour post dose: number analyzed (Participants) | 3 | 5 | 20
  Day 14: 72 hour post dose | 0.4900 (0.43025) | 1.070 (1.5187) | 0.8378 (0.72049)

14. Other Pre Specified Outcome: Plasma Concentration Versus Time Summary of Multiple Dose of OAP-189
Description: Concentration versus time summary was calculated by setting concentration values below the lower limit of quantification (LLOQ =0.500 nanogram per millliter) to zero. Summary statistics were not to be presented if number of observations above lower limit of quantification (NALQ) =0.
Time Frame: Pre-dose (2 hours before dosing), 1, 2, 3, 4, 6, 8, 10, 12, 14, 16, 24 hours post-dose on Day 7
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Arm/Group | OAP-189 0.2 mg IR | OAP-189 0.4 mg IR
Number analyzed (Participants) | 10 | 14
nanogram per milliliter
  Pre-dose | 1.667 (1.4404) | 3.548 (1.9612)
  1 hour post dose | 2.727 (1.4936) | 4.920 (1.7474)
  2 hour post dose | 4.454 (2.9789) | 7.824 (2.9187)
  3 hour post dose | 5.614 (3.0258) | 10.09 (3.9267)
  4 hour post dose | 6.080 (3.0045) | 11.79 (5.0857)
  6 hour post dose | 5.206 (2.0969) | 9.204 (4.3138)
  8 hour post dose | 4.064 (1.6576) | 6.889 (2.7902)
  10 hour post dose | 2.743 (1.0067) | 5.076 (2.0844)
  12 hour post dose | 5.315 (2.0278) | 9.376 (3.7875)
  14 hour post dose | 6.976 (2.7327) | 11.61 (6.2016)
  16 hour post dose | 6.157 (1.8865) | 10.87 (4.9706)
  24 hour post dose | 1.315 (0.87065) | 2.591 (1.3243)

ADVERSE EVENTS:
Arm/Group | OAP-189 0.2 mg IR | OAP-189 0.4 mg IR | OAP-189 MR (0.05:1 Z/P Ratio) 0.9 mg Followed by 1.2 mg | OAP-189 MR (0.1:1 Z/P Ratio) 1.2 mg Followed by 1.6 mg | OAP-189 MR (0.25:1 Z/P Ratio) 1.2 mg Followed by 1.6 mg | Placebo IR | Placebo MR
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/15 | 0/13 | 0/12 | 0/20 | 0/5 | 0/16
Other Adverse Events (participants affected / at risk) | 6/11 | 11/15 | 13/13 | 10/12 | 16/20 | 1/5 | 11/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OAP-189 0.2 mg IR (N=11) | OAP-189 0.4 mg IR (N=15) | OAP-189 MR (0.05:1 Z/P Ratio) 0.9 mg Followed by 1.2 mg (N=13) | OAP-189 MR (0.1:1 Z/P Ratio) 1.2 mg Followed by 1.6 mg (N=12) | OAP-189 MR (0.25:1 Z/P Ratio) 1.2 mg Followed by 1.6 mg (N=20) | Placebo IR (N=5) | Placebo MR (N=16)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 2 | 3 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 2 | 4 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 3 | 3 | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 3 | 2 | 2 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 1 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 5 | 0 | 2 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 2 | 3 | 2 | 0 | 0 | 2
Hyperchlorhydria (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 8 | 9 | 6 | 8 | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 8 | 2 | 5 | 4 | 0 | 2
Vomiting projectile (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Application site irritation (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Asthenia (General disorders) | 1 | 2 | 0 | 2 | 1 | 0 | 0
Chills (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Inflammation (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infusion site inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection site erythema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Injection site haematoma (General disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 1
Injection site pain (General disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sluggishness (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 3 | 3 | 4 | 2 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0
Polydipsia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 5 | 2 | 2 | 2 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 3 | 2 | 5 | 4 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 3
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 0 | 1 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Umbilical erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Data for fasting Insulin level abnormalities and capillary glucose level abnormalities was not reported due to change in planned analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.